CLINICAL TRIAL: NCT03381651
Title: Different Radiation Dose of Neoadjuvant Chemoradiation Followed by Surgery in Treating Patients with Locally Advanced, Resectable Thoracic Esophageal Cancer
Brief Title: Different Radiation Dose of Neoadjuvant Chemoradiation for Resectable Thoracic Esophageal Squamous Carcinoma
Acronym: Neo-DRATEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Qixun Chen, Director, Head of thoracic surgery, Zhejiang Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZhejiangEC5040
Record Dates: First submitted 2017-12-18; First posted 2017-12-22 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2022-03

CONDITIONS: Esophageal Carcinoma; Neoadjuvant Chemoradiotherapy; Surgery
Keywords: Radiation dose
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Higher dose (50.4Gy/28F) of neoadjuvant chemoradiation (Active Comparator): Neoadjuvant chemoradiation: RT: 50.4Gy/28F/5.6W; CT: paclitaxel 50mg/m2 d1, qw + CBP AUC2 d1, qw, weekly for 6 wks; Surgery: 4-6 weeks after nCRT
  Interventions: Radiation: Higher dose (50.4Gy/28F) of neoadjuvant chemoradiation
- Lower dose (41.4Gy/23F) of neoadjuvant chemoradiation (Active Comparator): Neoadjuvant chemoradiation: RT: 41.4Gy/23F/4.6W; CT: paclitaxel 50mg/m2 d1, qw + CBP AUC2 d1, qw, weekly for 5 wks; Surgery: 4-6 weeks after nCRT
  Interventions: Radiation: Lower dose (41.4Gy/23F) of neoadjuvant chemoradiation

INTERVENTIONS:
Radiation: Higher dose (50.4Gy/28F) of neoadjuvant chemoradiation — 50.4Gy/28F radiation and concurrent chemotherapy with paclitaxel plus CBP used weekly
  Arms: Higher dose (50.4Gy/28F) of neoadjuvant chemoradiation
Radiation: Lower dose (41.4Gy/23F) of neoadjuvant chemoradiation — 41.4Gy/23F radiation and concurrent chemotherapy with paclitaxel plus CBP used weekly
  Arms: Lower dose (41.4Gy/23F) of neoadjuvant chemoradiation

SUMMARY:
Esophageal cancer is one of the most common cancers worldwide, while more than half new cases and deaths occurred in China. Surgery is the main curative treatment for this disease, the 5-year survival of EC remains poor, since most diseases are diagnosed at advanced stages.

In last decades, several large clinical trials and meta-analyses have demonstrated that neo-adjuvant chemoradiotherapy followed by surgery can significantly increase the overall survival of patients with EC compared with surgery alone, while no effect of nCRT was apparent on postoperative health-related quality of life . However, the optimal radiation dose and surgery timing are still unknown.

The investigators hypothesize that patients who receive higher dose (50.4Gy/28F) of neoadjuvant chemoradiation will have better pathologic response and progress-free survival compared to lower dose (41.4Gy/23F) of chemoradiation followed by surgery.

ELIGIBILITY:
Inclusion Criteria:

Age:18-70 years

Histologically verified squamous carcinoma of the thoracic esophagus.

Patients with performance status 0-1 according to the Eastern Cooperative Oncology Group (ECOG) scale at the pre CRT evaluation and judges to be fit for surgery at the pre and post CRT evaluations.

Tumors should be resectable or potentially resectable and without distant metastasis, as assessed before neoadjuvant CRT, including clinical stage T2-4N0M0 or T1-4N1M0 according to the 6th AJCC system.

Joined the study voluntarily and signed informed consent form

No surgical contraindications

No serious system dysfunction and immuno-deficiency, Adequate organ function including the following: Hemoglobin ≥10 g/dL, Neutrophils (ANC )≥1.5x109/L, platelet count ≥100x 109/L, TBIL<1.5 x ULN, ALT and AST ≤ 2.5 x ULN, creatinine≤1.5 x ULN

Exclusion Criteria:

Cervical esophageal cancer (The upper end of the lesion is in the esophagus of the cervical segment).

Patients with biopsy (by endoscopic ultrasound, laparoscopy, or laparotomy) proven metastatic supraclavicular or celiac nodes are ineligible.

Invasion of the tracheobronchial tree or aorta

Tracheoesophageal fistula

Concurrent pregnancy or lactation

Severe diabetes mellitus with poor blood glucose control

History of a second malignancy

Patients being unable to undergo esophageal reconstruction with gastric tube, due to prior surgery.

Patients undergoing esophageal reconstruction with jejunum.

Patients have allergy reaction or contraindications to taxanes.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2018-02-22 (Actual); Primary Completion 2021-02-22 (Actual); Study Completion 2023-02-22 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 2 year
  Time from randomization to tumor progression or any deaths

SECONDARY OUTCOMES:
R0 resection rate in each arm | analysis is completed 4 weeks after surgery
  no cancer cells seen microscopically at the resection margin
Complete pathological response rate | analysis is completed 4 weeks after surgery
  using the Chirieac grading system
Postoperative complications in each study arm | 30 and 90 days after surgery
  According to the NCI CTC3.0
Treatment failure pattern | 2 year
  including local recurrence or distant metastasis or both
Overall survival | 5 year
  by intention to treat and per protocol analyses in each study arm

CONTACTS AND LOCATIONS:
Overall Officials: Weimin Mao, M.D., Principal Investigator — Zhejiang Caner Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sjoquist KM, Burmeister BH, Smithers BM, Zalcberg JR, Simes RJ, Barbour A, Gebski V; Australasian Gastro-Intestinal Trials Group. Survival after neoadjuvant chemotherapy or chemoradiotherapy for resectable oesophageal carcinoma: an updated meta-analysis. Lancet Oncol. 2011 Jul;12(7):681-92. doi: 10.1016/S1470-2045(11)70142-5. Epub 2011 Jun 16. PMID 21684205
- [Background] Shapiro J, van Lanschot JJB, Hulshof MCCM, van Hagen P, van Berge Henegouwen MI, Wijnhoven BPL, van Laarhoven HWM, Nieuwenhuijzen GAP, Hospers GAP, Bonenkamp JJ, Cuesta MA, Blaisse RJB, Busch ORC, Ten Kate FJW, Creemers GM, Punt CJA, Plukker JTM, Verheul HMW, Bilgen EJS, van Dekken H, van der Sangen MJC, Rozema T, Biermann K, Beukema JC, Piet AHM, van Rij CM, Reinders JG, Tilanus HW, Steyerberg EW, van der Gaast A; CROSS study group. Neoadjuvant chemoradiotherapy plus surgery versus surgery alone for oesophageal or junctional cancer (CROSS): long-term results of a randomised controlled trial. Lancet Oncol. 2015 Sep;16(9):1090-1098. doi: 10.1016/S1470-2045(15)00040-6. Epub 2015 Aug 5. PMID 26254683
- [Background] Tepper J, Krasna MJ, Niedzwiecki D, Hollis D, Reed CE, Goldberg R, Kiel K, Willett C, Sugarbaker D, Mayer R. Phase III trial of trimodality therapy with cisplatin, fluorouracil, radiotherapy, and surgery compared with surgery alone for esophageal cancer: CALGB 9781. J Clin Oncol. 2008 Mar 1;26(7):1086-92. doi: 10.1200/JCO.2007.12.9593. PMID 18309943
- [Background] Gebski V, Burmeister B, Smithers BM, Foo K, Zalcberg J, Simes J; Australasian Gastro-Intestinal Trials Group. Survival benefits from neoadjuvant chemoradiotherapy or chemotherapy in oesophageal carcinoma: a meta-analysis. Lancet Oncol. 2007 Mar;8(3):226-34. doi: 10.1016/S1470-2045(07)70039-6. PMID 17329193
- [Background] Noordman BJ, Verdam MGE, Lagarde SM, Hulshof MCCM, van Hagen P, van Berge Henegouwen MI, Wijnhoven BPL, van Laarhoven HWM, Nieuwenhuijzen GAP, Hospers GAP, Bonenkamp JJ, Cuesta MA, Blaisse RJB, Busch OR, Ten Kate FJW, Creemers GM, Punt CJA, Plukker JTM, Verheul HMW, Spillenaar Bilgen EJ, van Dekken H, van der Sangen MJC, Rozema T, Biermann K, Beukema JC, Piet AHM, van Rij CM, Reinders JG, Tilanus HW, Steyerberg EW, van der Gaast A, Sprangers MAG, van Lanschot JJB. Effect of Neoadjuvant Chemoradiotherapy on Health-Related Quality of Life in Esophageal or Junctional Cancer: Results From the Randomized CROSS Trial. J Clin Oncol. 2018 Jan 20;36(3):268-275. doi: 10.1200/JCO.2017.73.7718. Epub 2017 Nov 21. PMID 29161204
- [Background] van Hagen P, Hulshof MC, van Lanschot JJ, Steyerberg EW, van Berge Henegouwen MI, Wijnhoven BP, Richel DJ, Nieuwenhuijzen GA, Hospers GA, Bonenkamp JJ, Cuesta MA, Blaisse RJ, Busch OR, ten Kate FJ, Creemers GJ, Punt CJ, Plukker JT, Verheul HM, Spillenaar Bilgen EJ, van Dekken H, van der Sangen MJ, Rozema T, Biermann K, Beukema JC, Piet AH, van Rij CM, Reinders JG, Tilanus HW, van der Gaast A; CROSS Group. Preoperative chemoradiotherapy for esophageal or junctional cancer. N Engl J Med. 2012 May 31;366(22):2074-84. doi: 10.1056/NEJMoa1112088. PMID 22646630
- [Background] Teoh AY, Chiu PW, Yeung WK, Liu SY, Wong SK, Ng EK. Long-term survival outcomes after definitive chemoradiation versus surgery in patients with resectable squamous carcinoma of the esophagus: results from a randomized controlled trial. Ann Oncol. 2013 Jan;24(1):165-71. doi: 10.1093/annonc/mds206. Epub 2012 Aug 10. PMID 22887465